CLINICAL TRIAL: NCT06884397
Title: Implantation of an Endovascular Prosthesis for the Treatment of Abdominal Aortic Aneurysms: Use of a Machine Learning Model From CT Images to Predict Complications
Brief Title: Use of Artificial Intelligence to Predict Complications Following Abdominal Aortic Surgery
Acronym: AORTAPREDICT
Status: Recruiting | Type: Observational
Sponsor: Groupe Hospitalier de la Rochelle Ré Aunis (Other)
Collaborators: La Rochelle University (Unknown)
Responsible Party: Sponsor
Other Study IDs: P01045
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Abdominal Aortic Aneurysms (AAA)
Keywords: Aortic Aneurysm, Abdominal; Prostheses and Implants; Endoleak; Angiography, Computed Tomography; machine learning algorithm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Endoleak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patient treated for an abdominal aortic aneurysm: Indications for infrarenal abdominal aortic aneurysm (AAA) treatment with abdominal aortic endoprosthesis (AAE) were :
  * AAAs with greatest diameter > 50 mm for women and > 55 mm for men, or diameter increase of more than 5 mm in six months and 10 mm in 1 year.
  * A symptomatic or complicated AAA is treated regardless of size.
  * Despite the absence of conclusive data, a saccular AAA is considered high-risk due to its particular morphology and is proposed for treatment even if its greatest diameter is < 50 mm.
  Interventions: Procedure: Abdominal aortic endoprosthesis

INTERVENTIONS:
Procedure: Abdominal aortic endoprosthesis — An endoprosthesis consisting of a metal spring covered with an impermeable fabric is inserted through an artery and deployed inside the aorta.

SUMMARY:
Abdominal aortic aneurysm, a condition characterised by an increase in the diameter of the aorta, can be treated either surgically or endovascularly. In the latter, an endoprosthesis consisting of a metal spring covered with an impermeable fabric is inserted through an artery and deployed inside the aorta. This new method appears to be less invasive than surgery, but its long-term results are not yet fully understood. As a result, patients who have undergone this treatment are monitored by their surgeon to ensure that there is no endoleak. Several research teams have proposed analysing medical images to predict this risk of endoleak. Doctors are now trying to use artificial intelligence to automate the analysis of these images.

DETAILED DESCRIPTION:
The use of endoprostheses has revolutionized the therapeutic management of patients with thoracic and/or abdominal aortic aneurysms.

In France, the placement of abdominal aortic endoprosthesis (AAE) for treating infrarenal abdominal aortic aneurysm (AAA) follows the recommendations of the French National Authority for Health (HAS) from 2001, updated in 2009 in light of medical device developments and subsequent literature data (2000-2006). It specifically states that: "endovascular treatment is less invasive than surgical treatment, allowing for reduced 30-day morbidity rates for patients eligible for both surgery and endovascular treatment." Endovascular treatment can thus be offered to patients with normal surgical risk and favorable anatomical criteria, alongside surgical treatment, after informing the patient about the benefits and risks of both methods. The vast majority of patients with AAE require regular long-term follow-up, focusing on sac dimension and volume analysis and complication management. All patients must simultaneously receive optimal treatment for their vascular risk factors and comorbidities.

The updated recommendations can be summarized as follows:

* Indications for treating asymptomatic infrarenal AAAs: AAAs with greatest diameter > 50 mm or diameter increase of more than 5 mm in six months and 10 mm in 1 year.
* A symptomatic or complicated AAA is treated regardless of size.
* Despite the absence of conclusive data, a saccular AAA is considered high-risk due to its particular morphology and is proposed for treatment even if its greatest diameter is < 50 mm.

Since 2009, the number of endoprosthetic treatments has steadily increased at the expense of open procedures, although a medical-economic evaluation has questioned the efficiency of endovascular technique in patients eligible for both techniques. The long-term benefit in preventing mortality from AAA rupture remains unestablished (the mortality benefit difference is not maintained at 4 years), and even though most patients die from their comorbidities rather than their aneurysm, the first deaths from late rupture (beyond the fifth year of implantation) have appeared in long-term follow-up studies.

Concurrently, these studies have shown that nearly half of treated patients will require one or more additional procedures in subsequent years, and among treated patients:

* Only those showing aneurysmal sac shrinkage are considered cured.
* An average volume reduction of 3.2% would be sufficient to prevent endoleak occurrence.
* Conversely, a volume increase of more than 2% would be significantly associated with endoleak existence.

Endoleak is the most common complication after AAE placement, with incidence varying greatly depending on type and time elapsed since endoprosthesis placement. It is defined by blood circulation between the AAE and the arterial wall of the AAA. Five types of endoleak have been described according to anatomical, chronological, or physiological characteristics:

* Type I Endoleak: Ia) proximal anterograde peri-prosthetic flow due to endoprosthesis fixation failure, Ib) distal retrograde peri-prosthetic flow due to endoprosthesis fixation failure, Ic) iliac occluder seal failure,
* Type II Endoleak: retrograde flow from lumbar artery(ies) or inferior mesenteric artery feeding the aneurysmal sac: IIa) reperfusion through inferior mesenteric artery, IIb) reperfusion through lumbar artery(ies)
* Type III Endoleaks: IIIa) separation of modular endoprosthesis components, IIIb) fabric degradation. Endoleaks indicating early mechanical failure or premature fatigue of the endoprosthesis, potentially facilitated by AAA morphological changes, particularly its retraction
* Type IV Endoleaks: excessive endoprosthesis porosity. Generally early (<30 days post-implantation), initially described but now almost non-existent due to fabric improvements
* Type V Endoleak: residual hyperpressure in the aneurysmal sac without obvious cause (no individualized leak) associated with AAA size increase. It warrants thorough investigation for endoleak and may lead to explantation.

Several teams have proposed preoperative criteria to predict endoleak risk (preoperative inferior mesenteric artery patency, sac size), but without real evidence. Some teams propose preventive embolizations based on these criteria (pre- or during procedure).

The investigators propose to evaluate whether a machine learning algorithm can predict endoleak risk from initial CT scan images.

ELIGIBILITY:
Inclusion Criteria:

* Treated for an abdominal aortic aneurysm through endovascular prosthesis implantation

Exclusion Criteria:

* Underwent intraoperative embolization of the inferior mesenteric artery or aneurysmal sac
* Refuse the use of their data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient treated at La Rochelle Hospital Centre for an abdominal aortic aneurysm through endovascular prosthesis implantation
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of endoleaks following endograft implantation | From AAE placement to the end of the two-year follow-up
  Endoleak is the most common complication after AAE placement, with incidence varying greatly depending on type and time elapsed since endoprosthesis placement. It is defined by blood circulation between the AAE and the arterial wall of the AAA. Five types of endoleak have been described according to anatomical, chronological, or physiological characteristics.

SECONDARY OUTCOMES:
Number of embolizations | From AAE placement to the end of the two-year follow-up
  Minimally invasive treatment that blocks one or more blood vessels or abnormal vascular channels
Sac size | Two-year follow-up
  Normal aortic diameter varies with age, sex, and body habitus, but the average diameter of the adult human infrarenal aorta is approximately 2.0 cm. In most adults, an aortic diameter >3.0 cm is generally considered aneurysmal.
Number of serious adverse events | From AAE placement to the end of the two-year follow-up
  deaths, ruptures, endoleaks, limb occlusions, and reinterventions

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Franco, MD, Study Director — Groupe Hospitalier de la Rochelle Ré Aunis
Locations (1):
- Groupe Hospitalier de la Rochelle Ré Aunis, La Rochelle, France

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available with publication. A Digital Object Identifier will be used and Data will be available at www.recherche.data.gouv.fr
Supporting Information: Study Protocol
Time Frame: Data will be available immediately following publication.
Access Criteria: Researchers who provide a methodologically sound proposal will have access to the data.

REFERENCES:
- [Background] Samura M, Morikage N, Otsuka R, Mizoguchi T, Takeuchi Y, Nagase T, Harada T, Yamashita O, Suehiro K, Hamano K. Endovascular Aneurysm Repair With Inferior Mesenteric Artery Embolization for Preventing Type II Endoleak: A Prospective Randomized Controlled Trial. Ann Surg. 2020 Feb;271(2):238-244. doi: 10.1097/SLA.0000000000003299. PMID 30946077
- [Background] Gentsu T, Yamaguchi M, Sasaki K, Kawasaki R, Horinouchi H, Fukuda T, Miyamoto N, Mori T, Sakamoto N, Uotani K, Taniguchi T, Koda Y, Yamanaka K, Takahashi H, Okada K, Hayashi T, Watanabe T, Nomura Y, Matsushiro K, Ueshima E, Okada T, Sugimoto K, Murakami T. Side branch embolization before endovascular abdominal aortic aneurysm repair to prevent type II endoleak: A prospective multicenter study. Diagn Interv Imaging. 2024 Sep;105(9):326-335. doi: 10.1016/j.diii.2024.03.003. Epub 2024 Mar 19. PMID 38503637
- [Background] Tinelli G, D'Oria M, Sica S, Mani K, Rancic Z, Resch TA, Beccia F, Azizzadeh A, Da Volta Ferreira MM, Gargiulo M, Lepidi S, Tshomba Y, Oderich GS, Haulon S; SLIM F-U EVAR, Collaborative Study Group. The sac evolution imaging follow-up after endovascular aortic repair: An international expert opinion-based Delphi consensus study. J Vasc Surg. 2024 Sep;80(3):937-945. doi: 10.1016/j.jvs.2024.03.007. Epub 2024 Mar 8. PMID 38462062